CLINICAL TRIAL: NCT03360695
Title: Bridge: Proactive Psychiatry Consultation and Case Management for Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Risk Management Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kelly Edwards Irwin, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-396; 1K08CA230185-01 (NIH)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Cancer; Severe Major Depression; Schizophrenia; Bipolar Disorder; Lung Cancer; Breast Cancer; Head and Neck Cancer; Gastrointestinal Cancer
Keywords: Cancer Care; Major Depression and Cancer; Schizophrenia and Cancer; Bipolar Disorder and Cancer; Lung Cancer; Breast Cancer; Head and Neck Cancer; Gastrointestinal Cancer; Schizophrenia; Bipolar Disorder; Major Depression
MeSH Terms: conditions — Neoplasms; Depressive Disorder, Major; Schizophrenia; Bipolar Disorder; Lung Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: 1. A consensus panel of disease-specific oncologists who are blinded to intervention arm will review all patients at 24 weeks of care and evaluate for disruptions in cancer care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proactive Psychiatry Consultation (PPC) - PILOT (Experimental): Proactive Psychiatry Consultation and Case Management is:
  1. Patient-centered: Based on the patient's needs, the team aims to build a relationship, increase engagement, and promote continuity.
  2. Team-based: A psychiatrist and case manager identify goals for cancer treatment, assess psychiatric history and symptoms with a focus on impact on cancer care, collaborate with community-based clinicians and caregivers, and address barriers to care.
  3. Integrated into cancer care delivery: The psychiatry and oncology teams collaborate starting at cancer diagnosis to support patient through cancer treatment.
  4. Systematic: The team monitors psychiatric and cancer-related symptoms and cancer care delivery to measure progress toward goals and rapidly adjust treatment as needed.
  Interventions: Other: Proactive Psychiatry Consultation (PPC)
- Proactive Psychiatry Consultation (PPC) - Randomized Trial (Experimental): Proactive Psychiatry Consultation and Case Management is:
  1. Patient-centered: Based on the patient's needs, the team aims to build a relationship, increase engagement, and promote continuity.
  2. Team-based: A psychiatrist and case manager identify goals for cancer treatment, assess psychiatric history and symptoms with a focus on impact on cancer care, collaborate with community-based clinicians and caregivers, and address barriers to care.
  3. Integrated into cancer care delivery: The psychiatry and oncology teams collaborate starting at cancer diagnosis to support patient through cancer treatment.
  4. Systematic: The team monitors psychiatric and cancer-related symptoms and cancer care delivery to measure progress toward goals and rapidly adjust treatment as needed.
  Interventions: Other: Proactive Psychiatry Consultation (PPC)
- Enhanced Usual Care (EUC) - Randomized Trial (Active Comparator): Study staff will send a templated email to the treating oncologist at enrollment informing the oncologists of the psychiatric diagnosis and available psychosocial services. Study staff will also inform the patient and caregiver of available psychosocial services.
  Interventions: Other: Enhanced Usual Care (EUC)

INTERVENTIONS:
Other: Proactive Psychiatry Consultation (PPC) — Proactive Psychiatry Consultation and Case Management aims to improve communication among the patient, oncology team, and mental health clinicians, and increase engagement of family and community caregivers, which may help patients to receive the cancer care they need.
  Arms: Proactive Psychiatry Consultation (PPC) - PILOT; Proactive Psychiatry Consultation (PPC) - Randomized Trial
Other: Enhanced Usual Care (EUC) — At enrollment, study staff will inform the treating oncologist of the psychiatric diagnosis and will inform the oncologist, patient, and caregiver of available psychosocial services.
  Arms: Enhanced Usual Care (EUC) - Randomized Trial

SUMMARY:
The purpose of this research is to understand if it is helpful for patients with mental illness to be connected to a psychiatrist and case manager at the time of cancer diagnosis.

DETAILED DESCRIPTION:
It is challenging to cope with cancer. The investigators want to understand if it is helpful for patients with serious mental illness (SMI) to be connected to a psychiatrist and case manager when cancer is diagnosed. Many people with illnesses like major depression, schizophrenia and bipolar disorder face barriers to receiving high quality cancer care. It can be difficult to get to appointments, have many different doctors, and experience depression or worry. Better communication between the patient, the oncology team, and mental health providers may improve care. As for all patients, it is important for people with mental illness to have access to high quality cancer treatment that is patient-centered and coordinated. Having a case manager and psychiatrist at the cancer center who collaborates with the oncology team starting at cancer diagnosis may help patients to receive the cancer care that they need.

This study includes a single-arm open pilot (n=8) to pilot patient and caregiver measures and refine the intervention manual; a run-in period (n=6) to pilot the randomized trial procedures; and a randomized controlled trial (n=120) to compare the impact of the Bridge model with enhanced usual care on disruptions in cancer care.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age ≥ 18 years old; Value ______
* Verbal fluency in English
* Serious mental illness (Schizophrenia spectrum disorder, bipolar disorder, or major depressive disorder with prior psychiatric hospitalization) confirmed by study clinician at consent
* Invasive breast, lung, gastrointestinal, or head and neck cancer (suspected or confirmed Stage I-III, or Stage IV cancer that can be treated with curative intent according to judgment by the oncologist.)
* Medical, surgical, or radiation oncology consultation at MGH Cancer Center within the past 8 weeks or a referral placed to the MGH Cancer Center and planned or recommended follow-up

Patient Exclusion Criteria:

* Have cognitive impairment severe enough to interfere with completing brief study assessments or providing informed consent (and does not have a guardian who can provide consent)
* Recurrence of the same cancer type

Caregiver Participants

* Age ≥ 18 years old; Value ______
* Verbal fluency in English
* Identified or confirmed by the patient or guardian as a caregiver
* Caregiver may be a relative, friend, or community mental health staff upon whom the patient relies upon for support and who accompanies the patient to medical appointments
* The caregiver should either live with the patient or have in-person contact with the patient once per week (on average)
* Patient or guardian must provide permission to contact caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly E Irwin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Irwin KE, Callaway CA, Corveleyn AE, Pappano CR, Barry MJ, Tiersma KM, Nelson ZE, Fields LE, Pirl WF, Greer JA, Temel JS, Ryan DP, Nierenberg AA, Park ER. Study protocol for a randomized trial of bridge: Person-centered collaborative care for serious mental illness and cancer. Contemp Clin Trials. 2022 Dec;123:106975. doi: 10.1016/j.cct.2022.106975. Epub 2022 Oct 25. PMID 36307008

RESULTS

PARTICIPANT FLOW:
Groups:
- Proactive Psychiatry Consultation (PPC) - Randomized Trial: Proactive Psychiatry Consultation and Case Management is:
  1. Patient-centered: Based on the patient's needs, the team aims to build a relationship, increase engagement, and promote continuity.
  2. Team-based: A psychiatrist and case manager identify goals for cancer treatment, assess psychiatric history and symptoms with a focus on impact on cancer care, collaborate with community-based clinicians and caregivers, and address barriers to care.
  3. Integrated into cancer care delivery: The psychiatry and oncology teams collaborate starting at cancer diagnosis to support patient through cancer treatment.
  4. Systematic: The team monitors psychiatric and cancer-related symptoms and cancer care delivery to measure progress toward goals and rapidly adjust treatment as needed.
  Proactive Psychiatry Consultation (PPC): Proactive Psychiatry Consultation and Case Management aims to improve communication among the patient, oncology team, and mental health clinicians, and increase engagement of family and community caregivers, which may help patients to receive the cancer care they need.
- Enhanced Usual Care (EUC) - Randomized Trial: CAREGIVERS: Enrolled caregivers of patients randomized to Enhanced Usual Care (EUC) arm of Randomized Trial.
- Proactive Psychiatry Consultation (PPC) - Randomized Trial: CAREGIVERS: Enrolled caregivers of patients randomized to Proactive Psychiatry Consultation (PPC) arm of Randomized Trial.
Period: Overall Study
Arm/Group | Enhanced Usual Care (EUC) - Randomized Trial | Proactive Psychiatry Consultation (PPC) - Randomized Trial | Enhanced Usual Care (EUC) - Randomized Trial: CAREGIVERS | Proactive Psychiatry Consultation (PPC) - Randomized Trial: CAREGIVERS
Started | 60 | 60 | 32 | 33
Completed | 57 | 58 | 32 | 33
Not Completed | 3 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics data were collected from patients and caregivers
Groups:
- Enhanced Usual Care (EUC) - Randomized Trial - CAREGIVERS: Enrolled caregivers of patients randomized to Enhanced Usual Care (EUC) arm of Randomized Trial.
- Proactive Psychiatry Consultation (PPC) - Randomized Trial - CAREGIVERS: Enrolled caregivers of patients randomized to Proactive Psychiatry Consultation (PPC) arm of Randomized Trial.
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care (EUC) - Randomized Trial | Proactive Psychiatry Consultation (PPC) - Randomized Trial | Enhanced Usual Care (EUC) - Randomized Trial - CAREGIVERS | Proactive Psychiatry Consultation (PPC) - Randomized Trial - CAREGIVERS | Total
Number analyzed (Participants) | 60 | 60 | 32 | 33 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data collected for patients ONLY.
  years
    number analyzed (Participants) | 60 | 60 | 0 | 0 | 120
    (all) | 62.0 (13.2) | 60.6 (11.8) |  |  | 61.3 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 25 | 15 | 8 | 12 | 60
  Female | 33 | 45 | 24 | 21 | 123
  Fluid / Non-Binary | 1 | 0 | 0 | 0 | 1
  Missing | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 56 | 56 | 32 | 32 | 176
  Unknown or Not Reported | 3 | 2 | 0 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 1 | 3 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 55 | 50 | 28 | 31 | 164
  More than one race | 1 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 1 | 3 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 32 | 33 | 120
Caregiver Enrolled [Count of Participants; unit: Participants] — Population: Data collected for patients ONLY.
  Participants
    number analyzed (Participants) | 60 | 60 | 0 | 0 | 120
    No caregiver enrolled | 28 | 27 |  |  | 55
    Caregiver enrolled | 32 | 33 |  |  | 65
Cancer Diagnosis [Count of Participants; unit: Participants] — Population: Cancer diagnosis data collected for patients ONLY.
  Participants
    number analyzed (Participants) | 60 | 60 | 0 | 0 | 120
    Breast | 14 | 20 |  |  | 34
    Gastrointestinal | 20 | 10 |  |  | 30
    Head & Neck | 14 | 14 |  |  | 28
    Lung | 12 | 16 |  |  | 28
Severe Mental Illness Diagnosis [Count of Participants; unit: Participants] — Population: SMI data collected for patients ONLY.
  Participants
    number analyzed (Participants) | 60 | 60 | 0 | 0 | 120
    Bipolar Depression | 25 | 22 |  |  | 47
    Depression | 24 | 26 |  |  | 50
    Schiz Spectrum Disorder | 11 | 12 |  |  | 23
Psychiatrist [Count of Participants; unit: Participants] — Population: Data point collected for patients ONLY.
  Participants
    number analyzed (Participants) | 60 | 60 | 0 | 0 | 120
    No psychiatrist | 26 | 35 |  |  | 61
    Has psychiatrist | 34 | 25 |  |  | 59
Relationship to Patient [Count of Participants; unit: Participants] — Relationship of caregiver to patient. Population: Data point collected for caregivers ONLY.
  Participants
    number analyzed (Participants) | 0 | 0 | 32 | 33 | 65
    Married / Living as if married |  |  | 14 | 14 | 28
    Non-cohabitating relationship |  |  | 3 | 1 | 4
    Divorced / separated |  |  | 1 | 0 | 1
    Friend |  |  | 1 | 1 | 2
    Family member |  |  | 9 | 14 | 23
    Work with through community mental health |  |  | 4 | 2 | 6
    Other |  |  | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disruptions in Cancer Care
Description: The number of patients who experience clinically relevant disruptions in cancer care (e.g. delay to cancer diagnosis or treatment, deviation from stage-appropriate cancer treatment, or interruption in planned treatment).
Time Frame: 6 months from study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care (EUC) - Randomized Trial | Proactive Psychiatry Consultation (PPC) - Randomized Trial
Number analyzed (Participants) | 57 | 58
Participants
  Any Disruption | 37 | 48
  No Disruption | 20 | 10

2. Secondary Outcome: BPRS (24)
Description: Brief Psychiatric Rating Scale (BPRS) 24
  24-item instrument where the rater enters a number for each symptom. Each symptom construct is rated on a Likert scale from 1 (NOT PRESENT) - 7 (EXTREMELY SEVERE). The sum of all 24 items is then calculated to a maximum score of 168 (24X7=168). The minimum score is 24 and the maximum score is 168. The higher the score, the more psychiatrically impaired the patient is. Higher scores mean worse psychiatric symptoms.
Time Frame: Week 0, Week 12, Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care (EUC) - Randomized Trial | Proactive Psychiatry Consultation (PPC) - Randomized Trial
Number analyzed (Participants) | 57 | 58
score on a scale
  Week 0 | 46.51 (11.25) | 47.44 (13.76)
  Week 12 | 43.06 (12.71) | 44.96 (12.26)
  Week 24 | 46.1 (14.03) | 41.22 (10.31)

3. Secondary Outcome: PHQ-9
Description: Patient Health Questionnaire-9 is a 9-item instrument that measures patient depression where a score of 1-4 indicates minimal depression, 5-9 Mild depression, 10-14 Moderate depression, 15-19 Moderately severe depression, 20-27 Severe depression. The minimum score is 1 and the maximum score is 27.
Time Frame: Week 0, Week 6, Week 12, Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care (EUC) - Randomized Trial | Proactive Psychiatry Consultation (PPC) - Randomized Trial
Number analyzed (Participants) | 57 | 58
score on a scale
  Week 0 | 9.67 (6.02) | 9.09 (6.72)
  Week 6 | 9.60 (5.98) | 7.89 (5.43)
  Week 12 | 9.78 (6.25) | 7.72 (5.77)
  Week 24 | 8.05 (6.34) | 6.93 (5.50)

ADVERSE EVENTS:
Time Frame: The specific duration of time over which each participant was assessed is equal to an average of 24 weeks.
Description: Adverse Event data was not collected for caregivers.
Arm/Group | Enhanced Usual Care (EUC) - Randomized Trial | Proactive Psychiatry Consultation (PPC) - Randomized Trial
All-Cause Mortality (participants affected / at risk) | 6/57 | 4/58
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/58
Other Adverse Events (participants affected / at risk) | 0/57 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT03360695/Prot_SAP_ICF_000.pdf